CLINICAL TRIAL: NCT01908283
Title: Influence of Immunosuppressive Treatment on Immunological Response to Pneumococcal Conjugated Vaccine (PCV13) in Patients With Inflammatory Bowel Disease
Brief Title: Induction of Immunity Against Streptococcus Pneumoniae in Adults With Inflammatory Bowel Disease
Acronym: PCV13inSIBDCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klara M. Pósfay Barbe (Other)
Collaborators: Swiss IBD Cohort Study (Unknown)
Responsible Party: Sponsor-Investigator, Klara M. Pósfay Barbe, Klara M. Posfay-Barbe, MD, MS, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCV13 in SIBDCS; SIBDCS Project n° 2012-17 (Other: Swiss IBD Cohort Study number)
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient non immunosuppressed (Experimental): Group 1 : patient without immunosuppressive treatment
  Interventions: Biological: 13-valent pneumococcal conjugated vaccine (PCV13)
- Patient immunosuppressed (Experimental): Group 2 : patient with immunosuppressive treatment
  Interventions: Biological: 13-valent pneumococcal conjugated vaccine (PCV13)

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugated vaccine (PCV13) — Immunization with 1 dose of PCV13 (=0.5ml) intra-muscular
  Other Names: Streptococcus pneumoniae conjugated vaccine; PCV13 (Prevenar13®, Pfizer AG, Zurich); Swissmedic authorization number 60129

SUMMARY:
Patients with inflammatory bowel disease are at increased risk for infections due to their baseline disease and the subsequent immunocompromising regimen. Streptococcus pneumoniae (pneumococcus) has a high mortality and morbidity, particularly in immunosuppressed patients. A polysaccharide vaccine covering 23 different serotypes of pneumococcus (PPSV23) is currently recommended to immunocompromised patients to reduce their risk of invasive pneumococcal infections (such as bacteremia, meningitis, or pneumonia). Its immunogenicity is however limited, both in magnitude and duration, even in healthy individuals. Several studies have investigated the immunogenicity of PPSV23 in patients with IBD and have reported a marked inhibitory effect of immunosuppressive therapy on vaccine responses.

A pneumococcal conjugated vaccine (PCV) was originally developed to protect young children and demonstrated as highly effective and safe. PCV13 contains polysaccharides from thirteen different serotypes, conjugated to an inactivated diphtheria toxin, and has the capacity to induce both primary and memory responses. PCV also appears much more immunogenic than PPSV23 in immunocompromised pediatric and adult patients. Whether some therapeutic regimens may nevertheless prevent the induction of protective responses by PCV13 is yet unknown.

To date, no study has yet reported the immunogenicity / safety of PCV13 in adult IBD patients.

Study's objectives

* Primary objective: evaluate the immunogenicity and safety profile of PCV13 immunization in IBD patients
* Secondary objective: evaluate the relative influence of treatment and disease on immune responses to PCV13 immunization
* Tertiary objective: evaluate the immunity/vulnerability against vaccine-preventable diseases (VZV, measles) in the IBD cohort of Switzerland (optional, depending on funds)

DETAILED DESCRIPTION:
A. Inclusion:

Patients are eligible for this study if they are part of the SIBDCS and are followed in Switzerland in Geneva, Vaud, Neuchatel or Bern. Gastroenterologist will present the study to the patient during a routine follow-up visit. Inclusion will be cumulative, into 2 groups of 150 patients without (Group 1) or with (Group 2) immunosuppressive treatments.

B. Intervention

1. Vaccine history evaluation: A questionnaire will be filled at baseline including questions to establish patients' history of vaccine-preventable diseases and/or immunizations.
2. Serologic evaluation: Blood will be taken at inclusion for a baseline serological evaluation against pneumococcus. Antibody analyses will be performed using enzyme linked immunosorbent assays (ELISA) to quantify antigen-specific immunoglobulin G (IgG) antibodies. Serological evaluation against tetanus, measles and VZV could be performed through a study extension, depending on funds available.
3. Pneumococcal immunization: PCV13 (1 dose=0.5ml, intra-muscular) will be administrated during the same inclusion visit.

   Optional intervention (depending on available funds):
4. Additional missing immunizations could be identified by the study team on an individualized level, based on the patient's immunological record, and presence or absence of immunosuppression.

C. Assessment of effectiveness:

A second blood sampling will be scheduled 2 months (minimum 1, maximum 4) after PCV13 administration and will to assess vaccine response to PCV13.

D. Assessment of safety:

Vaccine safety will be monitored using standardized diary cards recording local and systemic side effects at week 1, 2, 4, 6, 8 after immunization. Patient will also be contacted by phone at week 6 by the investigator who will ask standardized questions regarding vaccine safety. Potential changes in disease activity (vaccine-induced flares) will be monitored during the following 6 months, through data collected in the SIBDCS database.

ELIGIBILITY:
Inclusion Criteria:

* Being part of the Swiss IBD Cohort Study
* Being followed in Geneva, Neuchatel, Vaud or Bern
* Adult >18 years-old
* informed consent form signed
* acceptance of PCV13 immunization

Exclusion Criteria:

* Current relapse defined as a Crohn's Disease Activity Index (CDAI) >150 for patients with Crohn's disease or a Modified Truelove-Witts Activity Index (MTWAI) >10 for patients with ulcerative colitis
* Actually pregnant or planned pregnancy in the next month
* Immunization with a pneumococcal vaccine (conjugated or polysaccharide) in the previous 5 years
* Previous severe systemic reaction to immunization (respiratory or circulative)
* Episode of fever in the last 24 hours

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
serologic response to PCV13 vaccine in patients with inflammatory bowel disease | 2 months after immunization
  Patients with inflammatory bowel disease will receive the PCV13 vaccine and a blood sample scheduled 2 months after will evaluate vaccine responses.

SECONDARY OUTCOMES:
safety of PCV13 administration in patients with inflammatory bowel disease | 6 months
  The safety of the PCV13 immunization in patient with inflammatory bowel disease will be evaluated using standardized side effect card, standardized phone call and data on disease disease activity via the SIBDCS database.
Evaluate the relative influence of treatment and disease on immune responses to PCV13 immunization | 2 months
  Mean pneumococcal antibody titers in Group 1 (patients without immunosuppressive treatments) and Group 2 (patients with immunosuppressive treatment) before and after immunization will be compared. Logistic regression will identify independent factor associated with seropositivity and magnitude of vaccine response.

CONTACTS AND LOCATIONS:
Overall Officials: Klara M. Posfay-Barbe, MD, MS, Principal Investigator — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Pittet LF, Verolet CM, Michetti P, Gaillard E, Girardin M, Juillerat P, Mottet C, Maillard MH, Siegrist CA, Posfay-Barbe KM; Swiss Inflammatory Bowel Disease Cohort Study Group. Risk of Vaccine-Preventable Infections in Swiss Adults with Inflammatory Bowel Disease. Digestion. 2021;102(6):956-964. doi: 10.1159/000516111. Epub 2021 May 10. PMID 33971650